CLINICAL TRIAL: NCT04195542
Title: Knowledge and Follow-up of Vitamin B9 Supplementation Recommendations for Women in the Periconceptional Period to Prevent Neural Tube Closure Defects: a Study Conducted With Health Professionnals and Women Who Have Just Given Birth in Rennes CHU.
Brief Title: Vitamin B9 Supplementation Recommendations in Rennes CHU
Acronym: QUALI B9
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_30032_QUALI B9
Record Dates: First submitted 2019-11-28; First posted 2019-12-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Spina Bifida or Spinal Dysraphism
Keywords: Spina Bifida; Spinal dysraphism; vitamin B9 supplementation; folic acid; neural tube closure defects; folate
MeSH Terms: conditions — Spinal Dysraphism | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women in obstetric ward in Rennes CHU: women in obstetric ward in Rennes CHU
  Interventions: Other: Questionnaire
- CHU professionals: All CHU professionals contacted via their email address
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — questionnaire assessing knowledge of the need to take vitamin B9 supplementation in women in the periconceptional period and the reasons why this supplementation is carried out or not

SUMMARY:
The study objective is to assess the knowledge and the follow-up of vitamin B9 supplementation recommendations for women in the periconceptional period to prevent neural tube closure defects. It will be conducted with health professionnals and women who have just given birth in Rennes CHU.

This study aimes to assess men's and women's knowledge of the need to take vitamin B9 supplementation in women in the periconceptional period and the reasons why this supplementation is carried out or not, in order to target our future prevention campaign.

This will allow comparing the results before and after the prevention campaign.

DETAILED DESCRIPTION:
Neural tube closure defects are among the most common birth defects. They are also called Spina Bifida or spinal dysraphism. According to the latest epidemiological studies in Europe based on the EUROCAT register (1991-2011), the prevalence of neural tube closure defects (including spinal dysraphisms as well as anencephaly and encephalocele) at birth is estimated at 9.105/10000 births in Europe (95% CI 8.94 to 9.27) and 12.02/10000 births in France.

The effectiveness of vitamin B9 (or folic acid or folate) supplementation in the periconceptional period on reducing the prevalence of neural tube closure defects has been widely demonstrated.

In France, the HAS (public health agency) recommends taking vitamin B9 between 1 month before and 2 months after conception, at a dose of 0.4 mg per day (5 mg per day in case of risk factors) since 2009. However, the proportion of women taking folic acid during periconceptional period is estimated at 1%.

The spina bifida - dysraphisms centre of the University Hospital Center of Rennes wishes to implement a campaign to prevent neural tube closure defects by supplementing with vitamin B9 during periconceptional period.

This study aimes to assess men's and women's knowledge of the need to take vitamin B9 supplementation in women in the periconceptional period and the reasons why this supplementation is carried out or not, in order to target our future prevention campaign.

This will allow comparing the results before and after the prevention campaign. Finally, such a study is an awareness-raising campaign by itself. The study objective is to assess the knowledge and the follow-up of vitamin B9 supplementation recommendations for women in the periconceptional period to prevent neural tube closure defects. It will be conducted with health professionnals and women who have just given birth in Rennes CHU.

A questionnaire will be administered to each study participant, among 2 distinct populations:

* Paper questionnaire for women who have just given birth during their stay in the maternity ward at the University Hospital of Rennes.
* Electronic questionnaire (Sphinx Déclic) sent to all CHU mailbox users.

ELIGIBILITY:
Inclusion Criteria:

Questionnaires to women who have just given birth:

* Women >= 18 years old, hospitalized in obstretric wards in Rennes CHU
* Having given birth within 2 weeks of completing the questionnaire

Questionnaires to hospital professionals:

* People working at the Rennes CHU
* Using a standard email address...@chu-rennes.fr

Exclusion Criteria:

Questionnaires to women who have just given birth:

* Non-French-speaking
* Cognitive impairment preventing understanding of the questionnaire and self-reporting
* Person under legal protection
* Person subject to a measure to safeguard justice
* Refusal to participate

Questionnaires to university hospital professionals:

- Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women in obstetric ward in Rennes CHU and All CHU professionals
Sampling Method: Non-Probability Sample
Enrollment: 1284 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
To assess the knowledge and the follow-up of vitamin B9 supplementation recommendations for women in the periconceptional period to prevent neural tube closure defects. | the inclusion day
  Proportion of people who were or had a spouse supplemented during her last pregnancy.

SECONDARY OUTCOMES:
To assess the proportion of people who are aware of the need for vitamin B9 supplementation during the periconceptional period. | the inclusion day
  Proportion of people who are aware of the need for vitamin B9 supplementation during the periconceptional period.
To describe the type of B9 vitamin supplementation taken by women before and during pregnancy (alone or in a multivitamin supplement) and the modalities of intake (dosage, frequency, duration before and during pregnancy, etc.) | the inclusion day
  Dosage, frequency, duration before and during pregnancy, type of supplementation alone or in a multivitamin supplement
To understand how respondents were informed of the value of this supplementation (through their studies, through a health professional, medias, their entourage…) | the inclusion day
  Source of information about supplementation (through their studies, through a health professional, medias, their entourage…)
To understand why women do not take any B9 supplementation : information not known, pregnancy not planned, refusal to take it despite a medical prescription, forgetfulness. | the inclusion day
  Reasons of take any B9 supplementation : information not known, pregnancy not planned, refusal to take it despite a medical prescription, forgetfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Emma BAJEUX, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU de Rennes, Rennes, France